CLINICAL TRIAL: NCT01270802
Title: A Randomized Controlled Pilot Trial Comparing Continued Antiretroviral Therapy With Tenofovir/Emtricitabine/Efavirenz (TDF/FTC/EFV) With Switch to Tenofovir/Emtricitabine/Raltegravir (TDF/FTC/RAL) on Changes in Endothelial Function and Markers of Bone Metabolism
Brief Title: Effects of Switching Efavirenz to Raltegravir on Vascular Function and Bone Markers in HIV-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Samir Gupta, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck 38258
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2013-10-24 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-11

CONDITIONS: HIV
Keywords: Endothelial function; Vitamin D; Efavirenz; Raltegravir
MeSH Terms: interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir/emtricitabine/efavirenz (Active Comparator): Tenofovir/emtricitabine/efavirenz
  Interventions: Drug: Tenofovir/emtricitabine/efavirenz
- Tenofovir/emtricitabine plus raltegravir (Experimental): Tenofovir/emtricitabine/efavirenz is switched to tenofovir/emtricitabine plus raltegravir
  Interventions: Drug: Tenofovir/emtricitabine; Drug: Raltegravir

INTERVENTIONS:
Drug: Tenofovir/emtricitabine — Efavirenz will be switched to raltegravir 400mg orally twice daily while continuing tenofovir/emtricitabine
  Other Names: Truvada
  Arms: Tenofovir/emtricitabine plus raltegravir
Drug: Tenofovir/emtricitabine/efavirenz — Continued therapy with tenofovir/emtricitabine/efavirenz
  Other Names: Atripla
  Arms: Tenofovir/emtricitabine/efavirenz
Drug: Raltegravir — Efavirenz will be switched to raltegravir 400mg orally twice daily while continuing tenofovir/emtricitabine
  Other Names: Isentress
  Arms: Tenofovir/emtricitabine plus raltegravir

SUMMARY:
Efavirenz, a commonly used HIV medication, may cause worsening vascular function and bone problems. The purpose of this study is to determine if switching efavirenz to raltegravir, a newer HIV medication, will improve vascular function and tests of bone health.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is an increasingly important comorbidity in HIV-infected patients. Our preliminary data suggests that efavirenz may worsen endothelial function, which in turn may increase the risk for future CVD events. Efavirenz has also been linked to lower vitamin D levels, which may in turn result in increased bone fragility. Raltegravir is not known to affect either endothelial function or vitamin D levels. Therefore, switching efavirenz to raltegravir in patients with suppressed HIV viremia may lead to improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by (1) any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or (2) by two detectable HIV-1 antigens, or (3) two detectable plasma HIV-1 RNA viral loads.
* Age equal to or greater than 18 years.
* Receipt of TDF/FTC/EFV as the subject's initial ART regimen for at least one year prior to Screening.

Note: Interruptions in TDF/FTC/EFV of up to 10 days total during the 90 days prior to screening are allowed.

Note: Subjects who had received 3TC (lamivudine) with TDF/EFV as part of their initial regimen but have received TDF/FTC/EFV for at least one year prior to screening will be eligible.

* HIV-1 RNA level <50copies/mL at screening and with a history of having an HIV-1 RNA level of <50copies/mL between 1 and 6 months prior to screening.
* At least one genotypic resistance test done prior to initiation of TDF/FTC/EFV suggesting no evidence of antiretroviral resistance to any nucleos(t)ide reverse transcriptase inhibitor or non-nucleoside reverse transcriptase inhibitor.
* No previous use of raltegravir or other integrase inhibitor.
* For women of reproductive potential, a negative urine pregnancy test at screening and willingness to use two forms of birth control during the course of the study. Acceptable forms of birth control include condoms (with or without a gel that can kill sperm), a diaphragm or cervical cap (with or without a gel that can kill sperm), an intrauterine device (IUD), or hormonal-based birth control ("the pill").

Exclusion Criteria:

* Inability to complete written, informed consent.
* Incarceration at the time of any study visit.
* Diagnosed vascular disease (history of angina pectoris, coronary disease, peripheral vascular disease, cerebrovascular disease, aortic aneurysm, or otherwise known atherosclerotic disease).
* Diagnosed disease or process, besides HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosis, inflammatory bowel diseases, other collagen vascular diseases).

Note: Hepatitis B or C co-infections are NOT exclusionary

* Known or suspected malignancy requiring systemic treatment within six months of screening.
* History of ADA-defined diabetes mellitus

Note: History of gestational diabetes is not exclusionary if the potential subject does not have current ADA-defined diabetes.

* History of migraine headaches.
* History of Raynaud's phenomenon.
* History of cardiac arrhythmias or cardiomyopathy.
* Uncontrolled hyperthyroidism or hypothyroidism, defined as TSH values outside of the local reference range on most recent clinical assessment.
* History of hypoparathyroidism or hyperparathyroidism, even if treated.
* Known allergy or intolerance to nitroglycerin.
* History of carotid bruits.
* Creatinine clearance < 50mL/min (using the Cockcroft-Gault equation) using a serum creatinine level measured at screening.
* Hemoglobin < 9.0mg/dL at screening.
* Alanine aminotransferase (ALT) level or aspartate aminotransferase (AST) > 3 times ULN at screening.
* Total bilirubin > 2.5 times ULN at screening.
* Fever, defined as T ≥ 38.0C within 48 hours prior to screening.

Note: Fever within 48 hours prior to each main study visit will require postponement of that study visit until the patient has defervesced (T < 38.0C) for at least 48 hours; fevers continuing past the allowed study visit timeframe will result in study discontinuation.

* Therapy for acute infection or other serious medical illnesses within 14 days prior to screening.

Note: Therapy for acute infection or other serious medical illnesses that overlaps with a main study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation.

* Pregnancy or breastfeeding during the course of the study.
* Hypotension, defined as systolic blood pressure < 90mmHg, at time of screening.

Note: Hypotension noted prior to brachial artery reactivity testing on each main study visit will result in study visit postponement of at least one day until systolic pressure is ≥ 90mmHg the morning of brachial reactivity testing; postponement outside of the allowed study visit timeframe will result in study discontinuation.

* Uncontrolled hypertension, defined as systolic blood pressure > 160mmHg or diastolic blood pressure > 100mgHg at screening.
* Receipt of investigational agents, cytotoxic chemotherapy, systemic glucocorticoids (of any dose), or anabolic steroids at screening.

Note: Physiologic testosterone replacement therapy is not exclusionary.

* Receipt of lipid-lowering drugs or anticonvulsants (defined as those drugs with significant CYP 450 induction or inhibition) screening.
* Use of sildenafil, vardenafil, or tadalafil within 72 hours (before or after) of each main study visit.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment into this trial occurred between April 2011 and May 2012. Participants were recruited from the HIV outpatient clinics associated with the Indiana University Health medical system.
Pre-assignment Details: Thirty-two persons screened for enrollment. Two of these failed screening (both for having screening HIV-1 RNA levels >50 copies/mL); the remaining 30 were equally randomized into the two study groups.
Groups:
- Continued Tenofovir/Emtricitabine/Efavirenz: Tenofovir/emtricitabine/efavirenz : Continued therapy with tenofovir/emtricitabine/efavirenz (as Atripla) one pill per day
- Switch to Tenofovir/Emtricitabine Plus Raltegravir: Tenofovir/emtricitabine/raltegravir : Tenofovir/emtricitabine/efavirenz (as Atripla one pill per day) will be switched to tenofovir/emtricitabine (as Truvada one pill per day) plus raltegravir (as Isentress) 400mg orally twice daily
Period: Overall Study
Arm/Group | Continued Tenofovir/Emtricitabine/Efavirenz | Switch to Tenofovir/Emtricitabine Plus Raltegravir
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Continued Tenofovir/Emtricitabine/Efavirenz: Tenofovir/emtricitabine/efavirenz : Continued therapy with tenofovir/emtricitabine/efavirenz
- Switch to Tenofovir/Emtricitabine/Raltegravir: Tenofovir/emtricitabine/efavirenz is switched to tenofovir/emtricitabine/raltegravir
  Tenofovir/emtricitabine/raltegravir : Efavirenz will be switched to raltegravir 400mg orally twice daily while continuing tenofovir/emtricitabine
- Total: Total of all reporting groups
Arm/Group | Continued Tenofovir/Emtricitabine/Efavirenz | Switch to Tenofovir/Emtricitabine/Raltegravir | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12) | 39 (10.6) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Dilation (FMD) of the Brachial Artery
Description: Change in FMD is a measure of change in endothelial function
Time Frame: Baseline and 24 weeks
Population: In the Switch to tenofovir/emtricitabine plus raltegravir arm, two FMD measurements at 24 weeks were removed from the analysis due to poor quality imaging.
Measure: Mean (Standard Deviation); unit: % change from baseline
Groups:
- Switch to Tenofovir/Emtricitabine Plus Raltegravir: Tenofovir/emtricitabine plus raltegravir 400mg orally twice daily
Arm/Group | Continued Tenofovir/Emtricitabine/Efavirenz | Switch to Tenofovir/Emtricitabine Plus Raltegravir
Number analyzed (Participants) | 13 | 12
% change from baseline | -0.67 (3.35) | -0.1 (3.26)
Statistical Analysis 1: Comparison: Continued Tenofovir/Emtricitabine/Efavirenz vs Switch to Tenofovir/Emtricitabine Plus Raltegravir; We assumed that the declines in FMD seen with TDF/FTC/EFV in our previous study would fully reverse. Thus, the clinically relevant effect size to be detected for FMD change was +3.12% (SD 4%) in those switching from EFV to RAL. Using a two-sample, independent, two-tailed t-test with 5% type I error and 20% type II error, a sample size of 13 per group would be needed to find a difference in FMD between groups. Allowing for a 10% dropout rate, we planned to recruit 15 subjects per group; Test type: Superiority or Other; p = 0.67, t-test, 2 sided — P-value was not adjusted for multiple comparisons; P<0.05 was considered statistically significant; Mean Difference (Net) = 0.81, 95% CI 2-sided [-0.75 to 2.37], Standard Error of Mean 0.76

2. Secondary Outcome: Change in Serum Levels of Vitamin D
Description: Change in serum levels of 24-OH-vitamin D provide a measure of the amount of change in vitamin D in the body
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Switch to Tenofovir/Emtricitabine Plus Raltegravir: Tenofovir/emtricitabine/efavirenz will be switched to tenofovir/emtricitabine plus raltegravir 400mg orally twice daily
Arm/Group | Continued Tenofovir/Emtricitabine/Efavirenz | Switch to Tenofovir/Emtricitabine Plus Raltegravir
Number analyzed (Participants) | 13 | 14
ng/mL | 0.06 (0.23) | 0.14 (0.25)
Statistical Analysis 1: Comparison: Continued Tenofovir/Emtricitabine/Efavirenz vs Switch to Tenofovir/Emtricitabine Plus Raltegravir; Test type: Superiority or Other; p = 0.40, t-test, 2 sided — P-value was not adjusted for multiple comparisons. P<0.05 was considered statistically significant; Mean Difference (Net) = -1.63, 95% CI 2-sided [-13.04 to 9.77], Standard Error of Mean 5.52

ADVERSE EVENTS:
Time Frame: 6 months
Description: Laboratory toxicities were assessed at week 8 and week 24.
Arm/Group | Continued Tenofovir/Emtricitabine/Efavirenz | Switch to Tenofovir/Emtricitabine/Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continued Tenofovir/Emtricitabine/Efavirenz (N=15) | Switch to Tenofovir/Emtricitabine/Raltegravir (N=15)
Virologic failure (Infections and infestations) | 1 (1) | 0 (0) — Confirmed HIV-1 RNA over 50 copies/mL
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Impaired fasting glucose (Endocrine disorders) | 1 (1) | 0 (0)
Diastolic hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was open-label. Correction for multiple testing was not performed, so apparently significant results may be falsely positive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No